CLINICAL TRIAL: NCT00516373
Title: A Phase I, Pharmacokinetic and Biological Evaluation of a Small Molecule Inhibitor of Poly ADP-Ribose Polymerase-1 (PARP-1), KU-0059436, in Patients With Advanced Tumours.
Brief Title: A Study to Assess the Safety and Pharmacokinetics of an Inhibitor of Poly ADP-Ribose Polymerase-1 (PARP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KU36-92; D0810C00002; 2005-001435-29 (EudraCT Number)
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Neoplasms; BRCA1 Protein; BRCA2 Protein
Keywords: advanced ovarian cancer; BRCA 1 protein; BRCA 2 protein; Poly(ADP ribose)polymerases
MeSH Terms: conditions — Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KU-0059436 (Experimental): KU-0059436 administered orally twice daily
  Interventions: Drug: KU-0059436 (AZD2281)(PARP inhibitor)

INTERVENTIONS:
Drug: KU-0059436 (AZD2281)(PARP inhibitor) — oral
  Other Names: Olaparib

SUMMARY:
To determine the safety, tolerability, dose-limiting toxicity (DLT), pharmacokinetic-pharmacodynamic profile, and maximum tolerated dose (MTD) of KU-0059436 when administered orally to patients with advanced solid tumours. To further evaluate the safety and efficacy of KU-0059436 in an expanded cohort of BCRA-enriched population, primarily ovarian cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Confirmed malignant advanced solid tumour refractory to standard therapy or for which no suitable effective standard therapy exists.

Exclusion Criteria:

* Anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the 4 weeks prior to trial entry (or a longer period depending on the defined characteristics of the agents used).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2005-07-11 (Actual); Primary Completion 2008-12-17 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, dose-limiting toxicity (DLT), and (MTD) of KU-0059436 | assessed at each visit

SECONDARY OUTCOMES:
Objective tumour response | assessed every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Dr. Johann De Bono, PhD MRCP FRCR, Principal Investigator — Royal Marsden Hospital Trust, London, UK
Locations (5):
- Research Site, Brussels, Belgium
- Research Site, Amsterdam, Netherlands
- Research Site, Szczecin, Poland
- United Kingdom (2):
  - Research Site, Edinburgh
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Matulonis UA, Penson RT, Domchek SM, Kaufman B, Shapira-Frommer R, Audeh MW, Kaye S, Molife LR, Gelmon KA, Robertson JD, Mann H, Ho TW, Coleman RL. Olaparib monotherapy in patients with advanced relapsed ovarian cancer and a germline BRCA1/2 mutation: a multistudy analysis of response rates and safety. Ann Oncol. 2016 Jun;27(6):1013-1019. doi: 10.1093/annonc/mdw133. Epub 2016 Mar 8. PMID 26961146
- [Derived] Ang JE, Gourley C, Powell CB, High H, Shapira-Frommer R, Castonguay V, De Greve J, Atkinson T, Yap TA, Sandhu S, Banerjee S, Chen LM, Friedlander ML, Kaufman B, Oza AM, Matulonis U, Barber LJ, Kozarewa I, Fenwick K, Assiotis I, Campbell J, Chen L, de Bono JS, Gore ME, Lord CJ, Ashworth A, Kaye SB. Efficacy of chemotherapy in BRCA1/2 mutation carrier ovarian cancer in the setting of PARP inhibitor resistance: a multi-institutional study. Clin Cancer Res. 2013 Oct 1;19(19):5485-93. doi: 10.1158/1078-0432.CCR-13-1262. Epub 2013 Aug 6. PMID 23922302
- [Derived] Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, Mortimer P, Swaisland H, Lau A, O'Connor MJ, Ashworth A, Carmichael J, Kaye SB, Schellens JH, de Bono JS. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009 Jul 9;361(2):123-34. doi: 10.1056/NEJMoa0900212. Epub 2009 Jun 24. PMID 19553641
- See also: CSR_Synopsis_D0810C00002(KU36-92).pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2678&filename=CSR_Synopsis_D0810C00002(KU36-92).pdf